CLINICAL TRIAL: NCT02011347
Title: Influence of Ketamine on a Closed-Loop Anesthesia System
Brief Title: Ketamine and Closed-Loop Anesthesia System
Acronym: LoopKeta
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012/26; 2012-003001-97 (EudraCT Number)
Record Dates: First submitted 2013-12-03; First posted 2013-12-13 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Anesthesia
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Patients will receive a closed-loop administration of propofol and remifentanil according to bispectral level and Ketamine (bolus dose of Ketamine (0.15 mg.kg-1) followed by an infusion of Ketamine (0.15 mg.kg-1 h-1) until the end of anesthesia)
  Interventions: Drug: Ketamine
- Placebo (Experimental): patients will receive a closed-loop administration of propofol and remifentanil according to bispectral level and a placebo (NaCl 9/00 (same volume as in the Ketamine group)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine
  Arms: Ketamine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective is to evaluate the sparing effect of ketamine on the dose of propofol.

ELIGIBILITY:
Inclusion Criteria:

* patients with an American Society of Anesthesiology score 1, 2 or 3
* scheduled for a surgical procedure lasting more than 2 hours under general anesthesia

Exclusion Criteria:

* pregnancy
* chronic pain
* simultaneous general and loco-regional anesthesia
* contra-indication to to nonsteroidal anti-inflammatory drug
* contra-indication to Ketamine
* contra-indication to propofol, to remifentanil, to morphine
* history of central nervous system disease
* patients receiving a psychotropic treatment
* patients with a pace-maker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10-07 (Actual); Study Completion 2015-10-07 (Actual)

PRIMARY OUTCOMES:
administered dose of propofol during maintenance of anesthesia | day 1

SECONDARY OUTCOMES:
bispectral index measurement | 1 day
  bispectral index modification due to ketamine infusion before induction of anesthesia
administered dose of propofol during induction of anesthesia | day 1
administered doses of remifentanil during induction and maintenance of anesthesia | day 1
delay (measured as minutes) between the end of propofol and remifentanil administration and the recovery from anesthesia | day 1
hemodynamic abnormalities requiring treatment | day 1
% of time with a bispectral index between 40 and 60 | day 1
postoperative morphine requirement | day 1
incidence of postoperative nausea and vomiting | day 1
White and Song score | day 1
% of patients with an explicit memorisation of the intraoperative period | second postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (2):
- France (2):
  - Hopital Foch, Suresnes, Hauts de Seine
  - Clinique Fontaine les Dijons, Fontaine-lès-Dijon